CLINICAL TRIAL: NCT01244152
Title: Lifestyle Improvement Through Food and Exercise (LIFE): Self-Management in African Americans With Diabetes and Hypertension
Brief Title: Self-Management in African Americans With Diabetes and Hypertension
Acronym: LIFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Elizabeth Lynch, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK074485-01A2
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Intensive diabetes self-management education
- Control Group (Active Comparator)
  Interventions: Behavioral: Enhanced standard diabetes education

INTERVENTIONS:
Behavioral: Intensive diabetes self-management education — 18 group classes led by a dietitian and peer supporters, and weekly telephone calls by peer supporters. Intervention focus was on diet and physical activity.
  Arms: Intervention
Behavioral: Enhanced standard diabetes education — 2 3-hour diabetes education classes taught by a health educator at a local clinic
  Arms: Control Group

SUMMARY:
The primary aim of the study is to design a group-based, culturally appropriate self-management skills training intervention for disadvantaged African-Americans with both diabetes and hypertension and to compile an intervention Manual of Operations (MOO). The investigators are developing an intervention to assist individuals in reducing weight and hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus (HgA1c>7%), requiring the patient to take at least one tablet per day or one insulin injection per day and a diagnosis of hypertension (130/80) requiring them to take at least one medication per day;
* Participants must identify themselves as African-American;
* Participant resides in or proximal to the North Lawndale neighborhood;
* Secure written permission from their physician to engage in moderate physical activity. This set of participants may be at high risk for cardiac disease and this exclusion avoids putting them at undue risk;
* BMI ≥ 25. Participant must be overweight because the main goal of our intervention is weight loss of 5% or more of initial body weight.

Exclusion Criteria:

* Diet-controlled diabetes;
* Hypertension controlled with lifestyle modification only;
* Endstage renal disease, stroke with paresis, congestive heart failure (NYHA class 3 or 4), or other major endorgan complication of diabetes;
* Comorbid conditions limiting probable life span to <4 years (e.g. cancer, AIDS) or indication of end-stage complications of diabetes (kidney dialysis, or transplant, blindness, or lower extremity amputation);
* Receiving treatment for a major psychiatric disorder (i.e. schizophrenia);
* Unable to give informed consent;
* Are under the age of 18-While type-2 diabetes and hypertension are increasing in those under the age of 18, adolescent medicine is a separate specialty area from adult medicine. Interventions should be targeted specifically toward this age group to take into consideration the specific emotional and psychological needs of adolescents;
* Alcoholism as measured by the CAGE.screener for alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Weight change

SECONDARY OUTCOMES:
Hemoglobin A1C

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lynch EB, Liebman R, Ventrelle J, Avery EF, Richardson D. A self-management intervention for African Americans with comorbid diabetes and hypertension: a pilot randomized controlled trial. Prev Chronic Dis. 2014 May 29;11:E90. doi: 10.5888/pcd11.130349. PMID 24874782